CLINICAL TRIAL: NCT01000922
Title: A Single Center, Randomized, Open-Label, Crossover Study, Comparing the Pharmacodynamic Properties of Insulin VIAJECT™, Regular Human Insulin, and Insulin Lispro Either in Combination With a Basal Insulin Infusion or With Insulin Glargine Relative to a Standardized Meal in Patients With Type 1 Diabetes
Brief Title: A Study Comparing the Pharmacodynamic Properties of Insulin VIAJECT™, Regular Human Insulin, and Insulin Lispro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biodel (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VIAJECT™-010JM
Record Dates: First submitted 2009-10-21; First posted 2009-10-23 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Diabetes Mellitus
Keywords: Mealtime Insulin; Rapid acting insulin; Ultra fast VIAject; prandial insulin
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Regular Human Insulin (Experimental): Single injection
  Interventions: Drug: Regular Human Insulin
- Lispro (Experimental): Single injection
  Interventions: Drug: Lispro
- VIAject (Experimental): Single injection
  Interventions: Drug: VIAject
- VIAject 50% (Experimental): Single injection
  Interventions: Drug: VIAject 50%
- VIAject/Insulin glargine (Experimental): Single injection
  Interventions: Drug: VIAject/Insulin Glargine
- Insulin Glargine/VIAject (Experimental): Single injection
  Interventions: Drug: Insulin Glargine/VIAject

INTERVENTIONS:
Drug: Regular Human Insulin — Individual dose of RHI administered subcutaneously
  Arms: Regular Human Insulin
Drug: Lispro — Individual dose of lispro administered subcutaneously
  Arms: Lispro
Drug: VIAject — Individual dose of VIAject administered subcutaneously
  Arms: VIAject
Drug: VIAject 50% — Individual dose of VIAject 50% administered subcutaneously
  Arms: VIAject 50%
Drug: VIAject/Insulin Glargine — VIAject mixed wiht insulin glargine and administered subcutaneously
  Arms: VIAject/Insulin glargine
Drug: Insulin Glargine/VIAject — Individual dose of VIAject and Insulin Glargine administered seperately and subcutaneously
  Arms: Insulin Glargine/VIAject

SUMMARY:
Evaluation of post-prandial blood glucose excursions after a standardized meal and pre meal injections of individual doses of the study insulins.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of type 1 diabetes for not less than 5 years
2. HbA1c values of not more than 9%
3. Age: 19 to 70 years
4. Sex: Male or Female
5. Body Mass Index: 18 - 28 kg/m2
6. Informed consent must be obtained in writing for all volunteers.

Exclusion Criteria:

1. Type 2 Diabetes mellitus.
2. History of hypersensitivity to any of the components in the study medication.
3. History of severe or multiple allergies.
4. Treatment with any other investigational drug in the last 1 month before study entry.
5. Treatment with any concomitant medication that in the judgment of the investigator. would interfere with the study results.
6. Progressive disease likely to prove fatal (e.g. malignancies).
7. Current drug or alcohol abuse, or a history which in the opinion of the Investigator will impair subject safety or protocol compliance.
8. Having a significant cardiovascular, respiratory, gastrointestinal, hepatic, renal, neurological, psychiatric and/or hematological disease as evaluated by the investigator.
9. Blood donation within the last 30 days.
10. A women who is lactating.
11. Pregnant women or women intending to become pregnant during the study.
12. A sexually active woman of childbearing age not actively practicing birth control by using a medically accepted device or therapy.
13. Positive Serology for HIV, Hepatitis B or Hepatitis C.
14. Abnormal ECG, safety lab or physical examination results that are deemed clinically significant by the investigator.
15. A lack of compliance or other reasons which, in the opinion of the investigator, prevent the participation of the subject in the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To compare the maximal post prandial blood glucose concentration and the time to maximal post prandial glucose concentration between the different treatments | 8 hours

SECONDARY OUTCOMES:
To compare the ppGlucmax for all treatments, the ppTGluc-max, the AUCGluc 0-180 and the AUCGluc 0-360, CGluc-baseline for all treatments. | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hompesch, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Profil Institute for Clinical Research, Inc. (PICR), Chula Vista, California, United States